CLINICAL TRIAL: NCT03192020
Title: DupuytrEn Treatment EffeCtiveness Trial (DETECT): Needle Fasciotomy, Surgery or Collagenase Injection for Dupuytren's Contracture
Brief Title: Trial Comparing Treatment Strategies in Dupuytren's Contracture
Acronym: DETECT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Central Finland Hospital District (Other); Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Tampere University Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Medcare Oy (Other); Finnish Institute for Health and Welfare (Other Government); Orton Orthopaedic Hospital (Other)
Responsible Party: Principal Investigator, Olli Leppänen, M.D., Ph.D., Tampere University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R17022M
Record Dates: First submitted 2017-06-08; First posted 2017-06-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Dupuytren Contracture
Keywords: Hand; Xiapex; Xiaflex; Clostridium histolyticum collagenase; Needle; Surgery; Aponeurectomy; Aponeurotomy; Fasciotomy; Fasciectomy; Dupuytren's disease; Dupuytren's contracture; Contracture; Connective tissue disease
MeSH Terms: conditions — Dupuytren Contracture; Contracture; Connective Tissue Diseases | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, outcome assessor blinded, three parallel armed (1:1:1), superiority trial comparing needle fasciotomy, collagenase injection and surgery as primary intervention for people with treatment-naïve Dupuytren's contracture with a five-year follow-up.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors who measured index, middle, ring and small fingers' flexion and extension degrees were blinded. Patients had opaque gloves in their hand when visiting the blinded outcome assessor. Due to the nature of the treatments it was not possible to blind patients, leading investigators or research assistants. To minimize any bias in interpreting the findings, we blinded treatment allocation in the draft results manuscript with groups labelled as A, B and C. The writing committee reached consensus on the interpretation of the findings prior to being unblinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Percutaneous needle fasciotomy (PNF) (Experimental): PNF is a treatment in which the Dupuytren's contracture cord causing the contracture is not excised, but only divided with a hypodermic needle.
  Interventions: Procedure: Percutaneous needle fasciotomy (PNF); Procedure: Limited fasciectomy (LF)
- Collagenase clostridium histolyticum (CCH) (Experimental): Generic name of the drug is collagenase clostridium histolyticum. Dosage form is injectable powder, dosage 0.58 mg and frequency is one injection in four weeks up to three times. One injection is performed normally at least to three different places in the cord.
  Interventions: Drug: Collagenase Clostridium Histolyticum (CCH) 2.9 MG/ML [Xiaflex]; Procedure: Limited fasciectomy (LF)
- Limited fasciectomy (LF) (Active Comparator): In LF, the thickened part of the palmar fascia causing the contracture is excised through skin incision.
  Interventions: Procedure: Limited fasciectomy (LF)

INTERVENTIONS:
Procedure: Percutaneous needle fasciotomy (PNF) — The division of the cord can be made under local anesthesia in the clinic and takes only a few minutes to perform. It can be performed whenever the cord is palpable. There are only puncture wounds left, and hence, the patient can start normal use of the hand the day after the procedure. If patient seeks for a treatment and the recurrence of the disease can not be treated by the PNF or patient is not willing to new PNF patient will be treated with LF.
  Other Names: Percutaneous needle aponeurotomy
  Arms: Percutaneous needle fasciotomy (PNF)
Drug: Collagenase Clostridium Histolyticum (CCH) 2.9 MG/ML [Xiaflex] — CCH chemically dissolves type I collagen of which the cord is composed of. It is injected inside the cord at least three different places in the outpatient clinic and the cord can be ruptured by gently force after one to three days. If patient seeks for a treatment and the recurrence of the disease can not be treated by the CCH or patient is not willing to new CCH patient will be treated with LF.
  Other Names: [Xiapex]
  Arms: Collagenase clostridium histolyticum (CCH)
Procedure: Limited fasciectomy (LF) — LF is performed in general or regional anesthesia in operating room. Constricting cords will be excised under direct vision. LF has been the dominant technique of surgical treatment. If patient seeks for a treatment the recurrence of the disease will be treated with LF as long as needed.
  Other Names: Limited aponeurectomy

SUMMARY:
Trial is a prospective, randomized, controlled, outcome assessor-blinded, three armed parallel 1:1:1, multicenter trial. The research objective is to determine, which treatment strategy 1) primary percutaneous needle fasciotomy (PNF) followed by surgical limited fasciectomy (LF) in patients who do not respond to PNF, 2) primary collagenase clostridium histolyticym (CCH) followed by LF in patients who do not respond to CCH or 3) LF as the primary (and secondary) treatment modality is the most cost-effective in treating Dupuytren´s contracture. Short- and long-term results will be published.

DETAILED DESCRIPTION:
Dupuytren's contracture (DC) is a fibroproliferative disorder of the palmar fascia, which in time leads to flexion contracture in one or more fingers. Etiology of the disease is still unknown, but it strongly seems that genetic factors play a major role. DC is associated most commonly with Caucasian population groups from Northern Europe. The estimated global prevalence among whites is 3% to 6% and increases with age. Men women ratio is 7:1. There is no definitive cure for DC. The treatment aims at relieving the symptoms by releasing the contracture by percutaneous or operative techniques.

The investigators planned a prospective, randomized, controlled, outcome assessor-blinded, three armed parallel 1:1:1, multicenter trial comparing the cost-effectiveness of 1) collagenase clostridium histolyticum followed by limited fasciectomy in non-responsive cases, 2) percutaneous needle fasciotomy followed by limited fasciectomy in non-responsive cases and 3) primary limited fasciectomy in short- and long-term follow-up in DC.

Protocol is approved by Tampere university hospital institutional review board and Finnish Medicine Agency (Fimea). All patients will give written informed consent. The results of the trial will be disseminated as published articles in peer-reviewed journals.

Treatment of Duputren's contracture aims at reducing the functional deficit caused by the contracture. Recurrence is almost inevitable if the follow-up is long enough. Therefore, the investigators aim to analyze the effectiveness of three different treatment strategies in long-term follow-up, in addition to short-term follow-up, which include multiple interventions rather than just single intervention. The investigators chose a pragmatic primary outcome, which comprises both objective and subjective standpoint and reflects the needs of the patients as well as goals of the healthcare system. Furthermore, our short-term results give good high quality level evidence of effectiveness of all the three treatments and long-term follow-up a good perspective to the cost-effectiveness of the strategies.

ELIGIBILITY:
Inclusion Criteria:

* patients with ≥20° passive extension deficit in metacarpophalangeal (MPJ) or proximal interphalangeal joint (PIPJ), or TPED ≥30° in MPJ and PIPJ of finger/fingers II-V
* age > 18 years
* palpable cord
* provision of informed consent
* ability to fill the Finnish versions of questionnaires.

Exclusion Criteria:

* recurrent contracture in the finger to be treated
* neurologic condition causing the loss of function of the finger to be treated
* contraindication for collagenase clostridium histolyticym (Xiapex/Xiaflex ®)
* pregnant or breast feeding
* total passive extension deficit > 135° (Tubiana stage 4) in finger to be treated
* rheumatoid arthritis
* previous fracture in finger to be treated, which affects range of motion of MPJ or PIPJ
* age > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of success | 5 year follow-ups
  Success is a composite outcome comprising of 1) at least 50% contracture release from the recruitment and 2) patient is in patient accepted symptom state (PASS). PASS is defined by question: "Would you be satisfied and not in need for any other treatment if the functional impairment caused by the contracture would remain the same as it is today for the rest of your life?". Primary time point is five years' follow-up visit.

SECONDARY OUTCOMES:
QuickDASH | 3 months, 2, 5 and 10 year follow-ups
  QuickDASH questionnaire is a validated upper extremity specific questionnaire consisting of 11 tasks/questions about the functional capacity and the pain.
Perceived hand function | 3 months, 2, 5 and 10 year follow-ups
  Perceived hand function will be assessed pre- and postoperatively by VAS scale.
Global rating | 3 months, 2, 5 and 10 year follow-ups
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better: This question is also used as anchor question in the MCII analysis in which +1 and +2 are considered to present meaningful improvement to the patient.
EQ-5D-3L | 3 months, 2, 5 and 10 year follow-ups
  EQ-5D-3L is a generic instrument for assessing quality of life comprising 5 dimensions and VAS for health level.
Rate of Patient Accepted Symptom State | 3 months, 2, 5 and 10 year follow-ups
  PASS is a relevant patient-centered outcome measurement, which reflects the overall state in which patients consider themselves as being well. It is a state of the symptoms between complete remission and subjective dissatisfaction with the symptoms.
Rate of patients achieving clinically significant improvement | 10 year follow-up
  Percentage of patients achieving clinically significant improvement (50% better PED) will be assessed.
Rate of patients achieving full contracture release | 3 months, 2, 5 and 10 year follow-ups
  Percentage of patients achieving full contracture release (PED 0°-5°) will be assessed.
Willingness to undergo same treatment | 3 months and 2 year follow-ups
  Patient satisfaction with the treatment will be assessed by a simple "yes" or "no" question: "Would you prefer the same treatment again, if the result would be the same as it is now?"
Major adverse events | 3 months, 2, 5 and 10 year follow-ups
  In the trial will be reported major adverse events, which include: tendon rupture, nerve injury, arterial injury, CRPS and infection, skin rupture or hematoma that needs hospitalization/revision surgery.
Extension deficits | 3 months, 2, 5 and 10 year follow-ups
  The total passive extension deficit (TPED) and passive extension deficit (PED) of metacarpophalangeal (MPJ) and proximal interphalangeal (PIPJ) joints are used in almost all of the DC studies. Most of the studies used the PED as their primary outcome. In this trial, the TPED and PED of MPJ and PIPJ are used as secondary outcomes.
Total maximum flexion | 3 months, 2, 5 and 10 year follow-ups
  Patients are seeking help for their extension deficit in DC but in the end flexion of the fingers is more important for the hand function. Our treatments should not jeopardize finger flexion in an effort to reduce the extension deficit.
Expenses | 2, 5 and 10 year follow-ups
  The costs are assessed by allocating previously estimated costs for interventions to each of the treatment arm.
Progression of the disease | 2, 5 and 10 year follow-ups
  Recurrence or extension is treated if the patient contacts the study center and requires new treatment (ie, patient is not in the PASS anymore) and at least 20° flexion contracture is observed in one of the joints. Progression of disease is measured and reported in three levels: (1) rate of reinterventions in the arm due to recurrence or extension of the disease (clinically relevant progression); (2) costs of reinterventions (impact of progression); and (3) change in TPED in those patients who do not require further treatments (clinically irrelevant progression).
Recurrence of the disease | 2, 5 and 10 year follow-ups
  In this study recurrence is defined when patient considers not being in PASS anymore and seeks for further treatment, and has at least 20° contracture.
Extension of the disease | 2, 5 and 10 year follow-ups
  Extension means that the disease will be activated in other rays than treated after the treatment.
Progression-free-survival | 2, 5 and 10 year follow-ups
  Progression-free-survival will be counted to each arm as mean time.
Favored treatment modality questionnaire | 2, 5 and 10 year follow-ups
  Favored treatment modality will be asked from patients who undergo several treatment modalities (i.e. LF after CCH or PNF). Outcome will be assessed by question: "If you presented with a contracture for the first time now, would you prefer needle fasciotomy/injectable drug as the primary treatment or would prefer having surgery at first place?"
Rate of success | 3 months, 2 and 10 year follow-ups
  Success is a composite outcome comprising of 1) at least 50% contracture release from the recruitment and 2) patient is in patient accepted symptom state (PASS). PASS is defined by question: "Would you be satisfied and not in need for any other treatment if the functional impairment caused by the contracture would remain the same as it is today for the rest of your life?". Primary time point is five years' follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mikko P Räisänen, M.D., Principal Investigator — Tampere University Hospital; Harry J Göransson, M.D., Ph.D., adjunct professor, Principal Investigator — Tampere University Hospital; Aleksi RP Reito, M.D., Ph.D., adjunct professor, Principal Investigator — Central Finland Central Hospital; Hannu Kautiainen, MSc, Principal Investigator — Medcare Ltd; Antti OV Malmivaara, M.D., Ph.D., adjunct professor, Principal Investigator — Finnish Institute for Health and Welfare
Locations (6):
- Finland (6):
  - Central Hospital of Central Finland, Jyväskylä, Central Finland
  - Oulu University hospital, Oulu, North Ostrobothnia
  - Kuopio University hospital, Kuopio, Northern Savonia
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University hospital, Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: Yes
All the IPD will be shared with other researchers by request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after finishing the trial and it will be available for 15 years.
Access Criteria: Request.

REFERENCES:
- [Background] Raisanen MP, Karjalainen T, Goransson H, Reito A, Kautiainen H, Malmivaara A, Leppanen OV. DupuytrEn Treatment EffeCtiveness Trial (DETECT): a protocol for prospective, randomised, controlled, outcome assessor-blinded, three-armed parallel 1:1:1, multicentre trial comparing the effectiveness and cost of collagenase clostridium histolyticum, percutaneous needle fasciotomy and limited fasciectomy as short-term and long-term treatment strategies in Dupuytren's contracture. BMJ Open. 2018 Mar 28;8(3):e019054. doi: 10.1136/bmjopen-2017-019054. PMID 29599391
- [Result] Raisanen MP, Leppanen OV, Soikkeli J, Reito A, Malmivaara A, Buchbinder R, Kautiainen H, Kaivorinne A, Stjernberg-Salmela S, Lappalainen M, Luokkala T, Ponkko A, Taskinen HS, Paakkonen M, Jaatinen K, Juurakko J, Karjalainen VL, Karjalainen T. Surgery, Needle Fasciotomy, or Collagenase Injection for Dupuytren Contracture : A Randomized Controlled Trial. Ann Intern Med. 2024 Mar;177(3):280-290. doi: 10.7326/M23-1485. Epub 2024 Feb 13. PMID 38346307
- Available data/document: Study Protocol — http://bmjopen.bmj.com/content/8/3/e019054 — Protocol in BMJ Open access

DOCUMENTS (1):
  • Informed Consent Form (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT03192020/ICF_001.pdf